CLINICAL TRIAL: NCT03284931
Title: A Randomized, Double-Blind, Multiple Dose, 3-way Crossover, Exploratory Study to Assess the Pharmacodynamic Effects of SAGE-217 Capsules in Healthy Adults Using a 5-hour Phase Advance Model of Insomnia
Brief Title: A Study to Assess the Pharmacodynamic Effects of SAGE-217 in Healthy Adults Using an Insomnia Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 217-EXM-101
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — zuranolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAGE-217 high dose (Experimental): SAGE-217
  Interventions: Drug: SAGE-217 high dose
- SAGE-217 low dose (Experimental): SAGE-217
  Interventions: Drug: SAGE-217 low dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAGE-217 high dose — high dose
  Arms: SAGE-217 high dose
Drug: Placebo — placebo
  Arms: Placebo
Drug: SAGE-217 low dose — low dose
  Arms: SAGE-217 low dose

SUMMARY:
This study will assess the pharmacodynamic effects of SAGE-217 in approximately 42 healthy adult subjects using an insomnia model.

DETAILED DESCRIPTION:
Subjects are expected to complete Treatment Periods 1, 2 and 3, followed by an optional open-label administration of SAGE-217 for pharmacokinetic purposes (Treatment Period 4).

This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to participate in the study, including all assessments, planned inpatient stays and all follow-up visits
* Subject is a healthy, ambulatory volunteer
* Subject meets sleep Qualification criteria

Exclusion Criteria:

* Subject has a medical history of suicidal behavior, epilepsy, eating disorders, sleep disorders, or circadian rhythm disorders
* Subject has worked a night shift or flown >1 time zone within 30 days prior to Screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency, as determined by polysomnography (PSG) | 16 days

SECONDARY OUTCOMES:
Safety and tolerability, as assessed by adverse events | 36 days
Safety and tolerability, as assessed by vital signs | 29 days
Safety and tolerability, as assessed by clinical laboratory data | 29 days
Safety and tolerability, as assessed by ECG | 29 days
Safety and tolerability, as assessed by Columbia Suicide Severity Rating Scale (C-SSRS) | 29 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sage Investigational Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/